CLINICAL TRIAL: NCT00979927
Title: A Placebo-controlled Double-blind, Randomised, Multiple Dose, Dose Escalating Study in Healthy Subjects to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SPC3649
Brief Title: SPC3649 Multiple Dose Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santaris Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPC3649-202; Eudract no 2009-012153-38
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Hepatitis C
Keywords: Antisense; miR-122 antagonist; safety in healthy Volunteers; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — miravirsen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Placebo Comparator)
  Interventions: Drug: saline
- SPC3649 (Active Comparator)
  Interventions: Drug: SPC3649

INTERVENTIONS:
Drug: SPC3649 — 5 weekly doses
  Arms: SPC3649
Drug: saline — 5 weekly doses
  Arms: Saline

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of SPC3649 given in multiple doses to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers: Males and postmenopausal females aged ≥ 18 to 60 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse events | Up to 169 Days

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of SPC3649 | Up to 169 Days
Effect on total Cholesterol | Up to 169 Days

CONTACTS AND LOCATIONS:
Overall Officials: Salah Hadi, MD,MSc, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA international, Zuidlaren, Netherlands